CLINICAL TRIAL: NCT06404437
Title: Detection of Aortic Stenosis With Smartphone Auscultation Using Machine Learning (HEARTBEAT-Pilot)
Status: Active, not recruiting | Type: Observational
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Collaborators: University of Erlangen-Nürnberg Medical School (Other); University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Johannes Michael Altstidl, Physician, Friedrich-Alexander-Universität Erlangen-Nürnberg
Other Study IDs: 23-39-B
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis
Keywords: Machine Learning; Digital Health; Heart Valve Disease; Cardiology
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases | interventions — Auscultation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe Aortic Stenosis
  Interventions: Diagnostic Test: Auscultation
- No Relevant Heart Valve Disease
  Interventions: Diagnostic Test: Auscultation

INTERVENTIONS:
Diagnostic Test: Auscultation — Auscultation at five auscultation points using a digital stethoscope and a smartphone

SUMMARY:
Severe aortic stenosis, a common heart valve issue, is usually treated surgically or through intervention. Diagnosis typically occurs after symptoms appear, but research suggests already treating asymptomatic cases may help patients live longer. Current diagnostics using echocardiography are detailed but time-consuming, prompting the exploration of a smartphone application using built-in microphones and machine learning for quicker and more accessible screening.

DETAILED DESCRIPTION:
Severe aortic stenoses usually is treated either surgically or interventionally, making it the most frequently treated among heart valve diseases. Typically, severe aortic stenosis is diagnosed only after the onset of the first symptoms. However, initial studies suggest that treating asymptomatic aortic stenoses could also extend the lifespan of affected individuals. Therefore, a widely applicable and cost-effective diagnostic method would be desirable for screening.

The current gold standard for diagnosing aortic stenosis is echocardiography. It allows for detailed measurement and evaluation, assisting in detection and diagnostic assessment. However, it is time-consuming and therefore not readily applicable to a larger population. Alternatively, auscultation as an acoustic method is suitable, where typical noise changes due to turbulence in blood flow can be detected using a stethoscope.

Since stethoscopes are only conditionally accessible for self-use, both in terms of availability and usability, this study aims to investigate whether a mobile application based on artificial intelligence for common smartphones using built-in microphones can also be diagnostically used. For this purpose, microphone recordings at the typical five auscultation points of 50 patients with severe aortic stenosis and 50 patients without any relevant heart valve disease are recorded. A digital stethoscope (3M Deutschland GmbH, Germany) and echocardiography findings serve as references. Based on the data, a classification model will be developed in a first step, which can detect severe aortic stenoses in smartphone recordings using machine learning.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* No relevant heart valve disease or severe aortic stenosis with no other relevant heart valve disease in echocardiography no older than 3 months

Exclusion Criteria:

* Previous surgerical or interventional therapy of a heart valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No relevant heart valve disease or severe aortic stenosis with no other relevant heart valve disease
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Algorithm Performance | Baseline
  Performance of algorithmic diagnosis measured by accuracy, sensitivity, specificity, and positive predictive value

SECONDARY OUTCOMES:
Comparison with Digital Stethoscope | Baseline
  Comparison of algorithm performance using smartphone recordings with algorithm performance using digital stethoscope recordings
Comparison of Auscultation Points | Baseline
  Comparison of algorithm performance using different sets of auscultation points

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Medicine 2 - Cardiology and Angiology, Friedrich-Alexander-Universität Erlangen-Nürnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Recordings and metadata are published
Supporting Information: Study Protocol, ICF, Analytic Code